CLINICAL TRIAL: NCT01106833
Title: A Phase II/III Randomized, Multicenter Trial Comparing Sirolimus Plus Prednisone and Sirolimus/Calcineurin Inhibitor Plus Prednisone for the Treatment of Chronic Graft-versus-Host Disease (BMT CTN Protocol #0801)
Brief Title: Chronic Graft-versus-Host Disease Treatment (BMT CTN 0801)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0801; U01HL069294 (NIH); BMT CTN 0801 (Other: Blood and Marrow Transplant Clinical Trials Network); U01HL06929406 (Other Grant/Funding Number: National Cancer Institute (NCI)); 5U24CA076518 (NIH)
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Chronic GVHD
Keywords: Chronic Graft-versus-Host Disease (cGVHD)
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Sirolimus; Calcineurin Inhibitors; Prednisone; Tacrolimus; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calcineurin inhibitor (Active Comparator): Sirolimus + calcineurin inhibitor + prednisone
  Interventions: Drug: Sirolimus + calcineurin inhibitor + prednisone
- Sirolimus and prednisone (Experimental): Sirolimus + prednisone
  Interventions: Drug: Sirolimus + prednisone

INTERVENTIONS:
Drug: Sirolimus + calcineurin inhibitor + prednisone — The target serum level for sirolimus is 3-12 ng/mL. The target serum level for tacrolimus is 5-10 ng/mL. The target serum level for cyclosporine is 120-200 ng/mL.
  Prednisone is administered initially as a single early morning dose of 1 mg/kg/day (or equivalent). If prednisone at a dose of 1 mg/kg/day (or equivalent) is contraindicated, patients may begin prednisone between 0.5-1 mg/kg/day.
  Other Names: Rapamune; Prograf; Neorall; Gengraf
  Arms: calcineurin inhibitor
Drug: Sirolimus + prednisone — The target serum level for sirolimus is 3-12 ng/mL.
  Prednisone is administered initially as a single early morning dose of 1 mg/kg/day (or equivalent). If prednisone at a dose of 1 mg/kg/day (or equivalent) is contraindicated, patients may begin prednisone between 0.5-1 mg/kg/day.
  Other Names: Rapamune
  Arms: Sirolimus and prednisone

SUMMARY:
This study is designed as a combined Phase II/III, randomized, open label, multicenter, prospective comparative study of sirolimus plus prednisone versus sirolimus/calcineurin-inhibitor plus prednisone for the treatment of chronic GVHD. Patients will be stratified by transplant center and will be randomized to an experimental arm of one of the two pre-specified experimental arms (sirolimus + prednisone or the comparator arm of sirolimus + calcineurin inhibitor + prednisone) in a 1:1 ratio.

DETAILED DESCRIPTION:
Background: Chronic GVHD is a medical condition that can become very serious. Chronic GVHD is a common development after allogeneic transplant that occurs when the donor cells attack and damage tissues. The primary purpose of this study is to compare treatment regimens that contain sirolimus without a calcineurin inhibitor to a comparator regimen of sirolimus with a calcineurin inhibitor and evaluate how well chronic GVHD responds to treatment. The combinations of medications in this study are:

* Sirolimus + calcineurin inhibitor + prednisone
* Sirolimus + prednisone

The goal is to select a treatment regimen for further comparison in the Phase III trial.

Design Narrative: The intent is to enroll subjects at the start of initial therapy for chronic GVHD, or before their chronic GVHD is refractory to glucocorticoid therapy, or is chronically dependent upon glucocorticoid therapy and multiple secondary systemic immunosuppressive agents. Patients will be stratified by transplant center and will be randomized to one of two arms.

ELIGIBILITY:
Inclusion Criteria:

* Suitable candidates are patients with classic chronic GVHD or overlap syndrome (classic chronic plus acute GVHD)that is: a)Previously untreated (newly diagnosed) as defined by having received < 14 days of prednisone (or equivalent) before enrollment/randomization to study therapy; b)Previously treated but inadequately responding after ≤ 16 weeks of initial therapy with prednisone and/or calcineurin inhibitor (CNI) ± additional non-sirolimus agent (started at the time of chronic GVHD diagnosis).
* Patient or guardian willing and able to provide informed consent.
* Stated willingness to use contraception in women of childbearing potential.
* Stated willingness of patient to comply with study procedures and reporting requirements.

Exclusion Criteria:

* Patients with late persistent acute GVHD or recurrent acute GVHD only.
* Inability to begin prednisone therapy at a dose of greater than 0.5 mg/kg/day.
* Receiving sirolimus for treatment of chronic GVHD (sirolimus for prophylaxis or treatment of acute GVHD is acceptable).
* Already receiving sirolimus (for prophylaxis or treatment of acute GVHD) with prednisone at ≥ 0.25 mg/kg/day (or equivalent) ± additional agents.
* Receiving therapy for chronic GVHD for more than 16 weeks.
* Invasive fungal or viral infection not responding to appropriate antifungal or antiviral therapies.
* Inadequate renal function defined as measured creatinine clearance less than 50 mL/min/1.73 m^2 based on the Cockcroft-Gault formula (adults) or Schwartz formula (age less than or equal to 12 years). Adults: estimated creatinine clearance rate (eCCr) (mL/min/) = (140 - age) x mass (kg) x (0.85 if female)/72 x serum creatinine (mg/dL; Creatinine clearance (mL/min/1.73m^2) = eCCr x 1.73/Body Surface Area (BSA) (m^2); Children: eCCr (mL/min/1.73 m^2) = k x height (cm) / serum creatinine (mg/dL) k = 0.33 (pre-term), 0.45 (full term to 1 year old), 0.55 (age 1-12 years).
* Inability to tolerate oral medications.
* Absolute neutrophil count less than 1500 per microliter.
* Requirement for platelet transfusions.
* Pregnancy (positive serum β-HCG) or breastfeeding.
* Receiving any treatment for persistent, progressive or recurrent malignancy.
* Progressive or recurrent malignancy defined other than by quantitative molecular assays.
* Known hypersensitivity to sirolimus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (31):
- United States (31):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Medical Center, La Jolla, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Blood & Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mayo Clinic, Rochester, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Jewish Hospital BMT Program, Cincinnati, Ohio
  - University Hospitals of Cleveland/ Case Western, Cleveland, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University (A) and (P), Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas/MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University/MCV Hospitals, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Derived] Carpenter PA, Logan BR, Lee SJ, Weisdorf DJ, Johnston L, Costa LJ, Kitko CL, Bolanos-Meade J, Sarantopoulos S, Alousi AM, Abhyankar S, Waller EK, Mendizabal A, Zhu J, O'Brien KA, Lazaryan A, Wu J, Nemecek ER, Pavletic SZ, Cutler CS, Horowitz MM, Arora M; BMT CTN.. A phase II/III randomized, multicenter trial of prednisone/sirolimus versus prednisone/ sirolimus/calcineurin inhibitor for the treatment of chronic graft-versus-host disease: BMT CTN 0801. Haematologica. 2018 Nov;103(11):1915-1924. doi: 10.3324/haematol.2018.195123. Epub 2018 Jun 28. PMID 29954931

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus, Calcineurin Inhibitor, and Prednisone: Sirolimus + calcineurin inhibitor + prednisone
  Sirolimus + calcineurin inhibitor + prednisone: The target serum level for sirolimus is 3-12 ng/mL.
  The target serum level for tacrolimus is 5-10 ng/mL. The target serum level for cyclosporine is 120-200 ng/mL.
  Prednisone is administered initially as a single early morning dose of 1 mg/kg/day (or equivalent). If prednisone at a dose of 1 mg/kg/day (or equivalent) is contraindicated, patients may begin prednisone between 0.5-1 mg/kg/day.
- Sirolimus and Prednisone: Sirolimus + prednisone
  Sirolimus + prednisone: The target serum level for sirolimus is 3-12 ng/mL.
  Prednisone is administered initially as a single early morning dose of 1 mg/kg/day (or equivalent). If prednisone at a dose of 1 mg/kg/day (or equivalent) is contraindicated, patients may begin prednisone between 0.5-1 mg/kg/day.
Period: Overall Study
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Started | 74 | 77
Completed | 74 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population includes only participants deemed to be eligible per Endpoint Review Committee adjudication. Thirteen enrolled participants were classified as ineligible (8 on the Sirolimus+Calcineurin Inhibitor+Prednisone arm and 5 on the Sirolimus+Prednisone arm) and are excluded from the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone | Total
Number analyzed (Participants) | 66 | 72 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (14.2) | 47.4 (16.1) | 49.1 (15.2)
Age, Customized [Count of Participants; unit: Participants] — Age in years
  Participants
    Less Than 20 | 2 | 5 | 7
    20 - 40 | 12 | 18 | 30
    41 - 60 | 36 | 30 | 66
    Over 60 | 16 | 19 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 24 | 57
  Male | 33 | 48 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 8
  Not Hispanic or Latino | 59 | 63 | 122
  Unknown or Not Reported | 7 | 1 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57 | 54 | 111
  Non-white | 9 | 13 | 22
  Unknown / Not Answered | 0 | 5 | 5
Primary Disease [Count of Participants; unit: Participants]
  Acute Leukemia | 25 | 47 | 72
  Chronic Leukemia | 8 | 7 | 15
  MDS / MPS | 9 | 12 | 21
  Lymphoma | 17 | 5 | 22
  Other | 7 | 1 | 8
Graft Type [Count of Participants; unit: Participants]
  Bone Marrow | 5 | 5 | 10
  Peripheral Blood Stem Cells | 60 | 64 | 124
  Single Cord Blood | 1 | 0 | 1
  Double Cord Blood | 0 | 3 | 3
Donor Type [Count of Participants; unit: Participants] — Population: Donor type is described only for bone marrow and peripheral blood cell transplants.
  Participants
    number analyzed (Participants) | 65 | 69 | 134
    Related | 38 | 29 | 67
    Unrelated | 27 | 40 | 67
Conditioning Regimen Intensity [Count of Participants; unit: Participants]
  Myeloablative | 29 | 47 | 76
  Non-myeloablative or Reduced Intensity | 37 | 25 | 62
Donor Age [Mean (Standard Deviation); unit: years] | 44.4 (15.2) | 38.5 (12.9) | 41.3 (14.0)
Donor Gender [Count of Participants; unit: Participants]
  Female | 26 | 35 | 61
  Male | 38 | 37 | 75
  Unknown | 2 | 0 | 2
Donor/Recipient Gender Matching [Count of Participants; unit: Participants]
  Female Donor, Female Recipient | 10 | 14 | 24
  Female Donor, Male Recipient | 16 | 21 | 37
  Male Donor, Female Recipient | 21 | 10 | 31
  Male Donor, Male Recipient | 17 | 27 | 44
  Unknown Donor Gender | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Treatment Success
Description: Treatment success was evaluated at 6 months in Phase II and is defined as a complete or partial response without secondary systemic immunosuppressive therapy and no recurrent malignancy or death. In Phase III, treatment success was evaluated at 24 months and is defined as a complete response without secondary systemic immunosuppressive therapy and no recurrent malignancy or death.
Time Frame: 6 months and 24 months post-randomization
Population: Twelve participants withdrew study consent between 6 and 24 months post-randomization, so are excluded from the analysis of treatment success at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
Participants
  Phase II: 6 Months: Yes | 33 | 35
  Phase II: 6 Months: No | 33 | 37
  Phase III: 24 Months: number analyzed (Participants) | 58 | 68
  Phase III: 24 Months: Yes | 9 | 10
  Phase III: 24 Months: No | 49 | 58
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportion of participants with treatment success at 6 months is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.63, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportion of participants with treatment success at 24 months is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.44, Fisher Exact — Two-sided testing was performed using a significance level of 0.05

2. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall survival is defined as survival of death from any cause.
Time Frame: 6 months and 24 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
percentage of participants
  6 Months | 85.5 [74.0 to 92.2] | 91.7 [82.4 to 96.2]
  24 Months | 74.0 [61.1 to 83.2] | 81.5 [70.3 to 88.8]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the rate of overall survival during the first two years post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.205, Log Rank — Two-sided testing was performed using a significance level of 0.05

3. Secondary Outcome: Percentage of Participants With Progression-free Survival
Description: Progression-free Survival is defined as survival without malignancy relapse. Relapse and death are considered failures for this endpoint.
Time Frame: 6 months and 24 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
percentage of participants
  6 Months | 84.0 [72.2 to 91.0] | 90.3 [80.7 to 95.2]
  24 Months | 67.3 [53.9 to 77.5] | 78.6 [67.1 to 86.5]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the rate of progression-free survival during the first two years post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.141, Log Rank — Two-sided testing was performed using a significance level of 0.05

4. Secondary Outcome: Percentage of Participants With Failure-free Survival
Description: Failure-free Survival is defined as survival without malignancy progression or initiation of secondary therapy for chronic GVHD. Progression, initiation of secondary therapy for chronic GVHD, and death are considered failures for this endpoint.
Time Frame: 6 months and 24 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
percentage of participants
  6 Months | 74.7 [62.3 to 81.4] | 73.6 [61.5 to 79.9]
  24 Months | 46.2 [33.4 to 58.1] | 48.6 [36.5 to 59.7]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the rate of failure-free survival during the first two years post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.775, Log Rank — Two-sided testing was performed using a significance level of 0.05

5. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse is defined as recurrence of the primary malignancy. Death is considered a competing risk for this endpoint.
Time Frame: 6 months and 24 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
percentage of participants
  6 Months | 4.8 [1.3 to 12.2] | 1.4 [0.1 to 6.7]
  24 Months | 14.9 [7.2 to 25.1] | 10.1 [4.4 to 18.6]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the rate of relapse during the first two years post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.396, Gray's test — Two-sided testing was performed using a significance level of 0.05; Death without relapse was treated as a competing risk

6. Secondary Outcome: Percentage of Participants With Secondary Immunosuppressive Therapy Initiated
Description: The percentage of participants initiating secondary immunosuppressive therapy for chronic GVHD is described. Death is considered a competing risk for this endpoint.
Time Frame: 6 months and 24 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
percentage of participants
  6 Months | 12.9 [6.0 to 22.5] | 13.9 [7.1 to 23.0]
  24 months | 29.4 [18.5 to 41.2] | 38.5 [27.1 to 49.8]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the rate of initiation of secondary immunosuppressive therapy for chronic GVHD during the first two years post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.219, Gray's test — Two-sided testing was performed using a significance level of 0.05; Death without initiation of secondary therapy is considered a competing risk for this endpoint

7. Secondary Outcome: Percentage of Participants With Discontinuation of Systemic Immunosuppressive Therapy at Two Years
Description: The percentage of participants discontinuing all systemic immunosuppressive therapy by two years post-randomization is described. Death is considered a competing risk for this endpoint.
Time Frame: 2 years post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
percentage of participants | 20 [10.9 to 31.0] | 23.2 [14.0 to 33.8]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the rate of discontinuation of systemic immunosuppressive therapy during the first two years post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.706, Gray's test — Two-sided testing was performed using a significance level of 0.05; Death without discontinuation of systemic immunosuppressive therapy is considered a competing risk for this endpoint

8. Secondary Outcome: Prednisone Dose
Description: Daily dose of prednisone is described by treatment arm at baseline, 6 months, and 1 year post-randomization.
Time Frame: Baseline, 6 months, and 1 year post-randomization
Population: Outcomes are analyzed in participants that were alive and completed assessments.
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
mg/kg/day
  Baseline: number analyzed (Participants) | 64 | 72
  Baseline | 0.9 [0.2 to 1.2] | 0.9 [0.2 to 2.1]
  6 Months: number analyzed (Participants) | 42 | 58
  6 Months | 0.2 [0.0 to 1.1] | 0.2 [0.0 to 0.8]
  1 Year: number analyzed (Participants) | 23 | 41
  1 Year | 0.2 [0.0 to 1.8] | 0.1 [0.0 to 0.9]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median prednisone dose at baseline is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.127, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median prednisone dose at 6 months post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.562, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 3: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median prednisone dose at 1 year post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.129, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05

9. Secondary Outcome: Change in Prednisone Dose From Baseline
Description: Change in the daily dose of prednisone from baseline, the time of randomization, is described by treatment arm at 6 months and 1 year post-randomization.
Time Frame: 6 months and 1 year post-randomization
Population: Outcomes are analyzed in participants that were alive and completed assessments.
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
mg/kg/day
  6 Months: number analyzed (Participants) | 42 | 58
  6 Months | -0.6 [-1.1 to 0.3] | -0.6 [-1.7 to 0.2]
  1 Year: number analyzed (Participants) | 23 | 41
  1 Year | -0.6 [-1.0 to 0.8] | -0.7 [-1.9 to -0.1]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median change in prednisone dose from baseline to 6 months post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.586, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median change in prednisone dose from baseline to 1 year post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.140, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05

10. Secondary Outcome: Serum Creatinine Level
Description: Creatinine level is described by treatment arm at baseline, 6 months, and 1 year post-randomization.
Time Frame: Baseline, 6 months, and 1 year post-randomization
Population: Outcomes are analyzed in participants that were alive and completed assessments.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
mg/dL
  Baseline | 0.9 [0.3 to 1.8] | 0.9 [0.4 to 1.6]
  6 Months: number analyzed (Participants) | 50 | 64
  6 Months | 1.0 [0.4 to 2.6] | 1.0 [0.5 to 1.6]
  1 Year: number analyzed (Participants) | 47 | 59
  1 Year | 0.9 [0.4 to 2.4] | 0.9 [0.4 to 1.7]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median serum creatinine level at baseline is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.582, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median serum creatinine level at 6 months post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.208, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 3: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median serum creatinine level at 1 year post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.431, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05

11. Secondary Outcome: Change in Serum Creatinine Level From Baseline
Description: Change in creatinine level from baseline, the time of randomization, is described by treatment arm at 6 months and 1 year post-randomization.
Time Frame: 6 months and 1 year post-randomization
Population: Outcomes are analyzed in participants that were alive and completed assessments.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
mg/dL
  6 Months: number analyzed (Participants) | 50 | 64
  6 Months | 0.1 [-0.8 to 1.8] | 0.1 [-0.6 to 1.1]
  1 Year: number analyzed (Participants) | 47 | 59
  1 Year | 0.0 [-0.5 to 1.2] | 0.0 [-0.5 to 0.6]
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median change in serum creatinine level from baseline to 6 months post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.147, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the median change in serum creatinine level from baseline to 1 year post-randomization is equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.863, Kruskal-Wallis — Two-sided testing was performed using a significance level of 0.05

12. Secondary Outcome: Patient-reported Chronic GVHD Severity
Description: Each patient's perception of the severity of the chronic GVHD was collected at baseline and at 6 months, 1 year, and 2 years post-randomization. Severity is categorized as none, mild, moderate, and severe.
Time Frame: Baseline, 6 months, 1 year, and 2 years post-randomization
Population: Outcomes are analyzed in participants that were alive and completed assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
Participants
  Baseline: number analyzed (Participants) | 54 | 62
  Baseline: None | 0 | 0
  Baseline: Mild | 21 | 20
  Baseline: Moderate | 23 | 32
  Baseline: Severe | 10 | 10
  Baseline: Relapsed | 0 | 0
  Baseline: Initiated Secondary Therapy | 0 | 0
  Baseline: Dead | 0 | 0
  6 Months: number analyzed (Participants) | 50 | 63
  6 Months: None | 4 | 6
  6 Months: Mild | 13 | 25
  6 Months: Moderate | 15 | 10
  6 Months: Severe | 2 | 3
  6 Months: Relapsed | 3 | 1
  6 Months: Initiated Secondary Therapy | 7 | 14
  6 Months: Dead | 6 | 4
  1 Year: number analyzed (Participants) | 53 | 60
  1 Year: None | 9 | 2
  1 Year: Mild | 13 | 23
  1 Year: Moderate | 4 | 3
  1 Year: Severe | 0 | 4
  1 Year: Relapsed | 5 | 3
  1 Year: Initiated Secondary Therapy | 15 | 21
  1 Year: Dead | 7 | 4
  2 Years: number analyzed (Participants) | 47 | 57
  2 Years: None | 2 | 6
  2 Years: Mild | 10 | 13
  2 Years: Moderate | 2 | 1
  2 Years: Severe | 0 | 0
  2 Years: Relapsed | 8 | 5
  2 Years: Initiated Secondary Therapy | 18 | 28
  2 Years: Dead | 7 | 4
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the patient-reported severity and vital status categories considered at baseline are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.620, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the patient-reported severity and vital status categories considered at 6 months post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.258, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 3: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the patient-reported severity and vital status categories considered at 1 year post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.036, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 4: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the patient-reported severity and vital status categories considered at 2 years post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.369, Fisher Exact — Two-sided testing was performed using a significance level of 0.05

13. Secondary Outcome: Provider-reported Chronic GVHD Severity
Description: Each patient's care provider's perception of the severity of the chronic GVHD was collected at baseline and at 6 months, 1 year, and 2 years post-randomization. Severity is categorized as none, mild, moderate, and severe.
Time Frame: Baseline, 6 months, 1 year, and 2 years post-randomization
Population: Outcomes are analyzed in participants that were alive and whose providers completed assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
Participants
  Baseline: number analyzed (Participants) | 63 | 72
  Baseline: None | 1 | 0
  Baseline: Mild | 13 | 17
  Baseline: Moderate | 46 | 48
  Baseline: Severe | 3 | 7
  Baseline: Relapsed | 0 | 0
  Baseline: Initiated Secondary Therapy | 0 | 0
  Baseline: Dead | 0 | 0
  6 Months: number analyzed (Participants) | 59 | 67
  6 Months: None | 6 | 2
  6 Months: Mild | 27 | 33
  6 Months: Moderate | 10 | 13
  6 Months: Severe | 0 | 0
  6 Months: Relapsed | 3 | 1
  6 Months: Initiated Secondary Therapy | 7 | 14
  6 Months: Dead | 6 | 4
  1 Year: number analyzed (Participants) | 56 | 64
  1 Year: None | 8 | 7
  1 Year: Mild | 15 | 19
  1 Year: Moderate | 5 | 9
  1 Year: Severe | 1 | 1
  1 Year: Relapsed | 5 | 3
  1 Year: Initiated Secondary Therapy | 15 | 21
  1 Year: Dead | 7 | 4
  2 Years: number analyzed (Participants) | 51 | 59
  2 Years: None | 7 | 7
  2 Years: Mild | 10 | 11
  2 Years: Moderate | 1 | 4
  2 Years: Severe | 0 | 0
  2 Years: Relapsed | 8 | 5
  2 Years: Initiated Secondary Therapy | 18 | 28
  2 Years: Dead | 7 | 4
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the provider-reported severity and vital status categories considered at baseline are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.450, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the provider-reported severity and vital status categories considered at 6 months post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.301, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 3: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the provider-reported severity and vital status categories considered at 1 year post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.750, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 4: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the provider-reported severity and vital status categories considered at 2 years post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.444, Fisher Exact — Two-sided testing was performed using a significance level of 0.05

14. Secondary Outcome: NIH Consensus Criteria Chronic GVHD Severity
Description: Chronic GVHD severity was determined at baseline and at 6 months, 1 year, and 2 years post-randomization per the 2005 NIH Consensus Criteria (Filipovich et al. 2005). Severity is categorized as none, mild, moderate, and severe.
Time Frame: Baseline, 6 months, 1 year, and 2 years post-randomization
Population: Outcomes are analyzed in participants that were alive and whose clinical assessments were completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
Participants
  Baseline: number analyzed (Participants) | 63 | 71
  Baseline: None | 0 | 1
  Baseline: Mild | 1 | 1
  Baseline: Moderate | 29 | 23
  Baseline: Severe | 33 | 46
  Baseline: Relapsed | 0 | 0
  Baseline: Initiated Secondary Therapy | 0 | 0
  Baseline: Dead | 0 | 0
  6 Months: number analyzed (Participants) | 59 | 67
  6 Months: None | 3 | 1
  6 Months: Mild | 3 | 3
  6 Months: Moderate | 25 | 27
  6 Months: Severe | 12 | 17
  6 Months: Relapsed | 3 | 1
  6 Months: Initiated Secondary Therapy | 7 | 14
  6 Months: Dead | 6 | 4
  1 Year: number analyzed (Participants) | 56 | 62
  1 Year: None | 2 | 3
  1 Year: Mild | 2 | 5
  1 Year: Moderate | 16 | 16
  1 Year: Severe | 9 | 10
  1 Year: Relapsed | 5 | 3
  1 Year: Initiated Secondary Therapy | 15 | 21
  1 Year: Dead | 7 | 4
  2 Years: number analyzed (Participants) | 58 | 68
  2 Years: None | 9 | 9
  2 Years: Mild | 6 | 12
  2 Years: Moderate | 8 | 8
  2 Years: Severe | 2 | 2
  2 Years: Relapsed | 8 | 5
  2 Years: Initiated Secondary Therapy | 18 | 28
  2 Years: Dead | 7 | 4
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the NIH Consensus Criteria severity and vital status categories considered at baseline are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.238, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the NIH Consensus Criteria severity and vital status categories considered at 6 months post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.546, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 3: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the NIH Consensus Criteria severity and vital status categories considered at 1 year post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.756, Fisher Exact — Two-sided testing was performed using a significance level of 0.05
Statistical Analysis 4: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the proportions of patients in the NIH Consensus Criteria severity and vital status categories considered at 2 years post-randomization are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.554, Fisher Exact — Two-sided testing was performed using a significance level of 0.05

15. Secondary Outcome: SF-36 Physical Component Summary
Description: The Medical Outcome Study SF-36 Physical Component Summary (PCS) is a subscale of the SF-36 intended to measure physical well-being. It is scored on a scale of 0-100, with higher scores indicating higher levels of well-being.
Time Frame: Baseline, 2 months, 6 months, 1 year, and 2 years post-randomization
Population: Outcomes are analyzed in participants that were alive and completed assessments.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
score on a scale
  Baseline: number analyzed (Participants) | 54 | 61
  Baseline | 38 (1.3) | 38 (1.2)
  2 Months: number analyzed (Participants) | 47 | 52
  2 Months | 39 (1.6) | 42 (1.6)
  6 Months: number analyzed (Participants) | 38 | 48
  6 Months | 38 (2.1) | 43 (1.5)
  1 Year: number analyzed (Participants) | 34 | 42
  1 Year | 40 (1.8) | 43 (1.7)
  2 Years: number analyzed (Participants) | 19 | 31
  2 Years | 44 (2.4) | 43 (2.0)
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean PCS scores at baseline are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.685, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean PCS scores at 2 months are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.105, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 3: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean PCS scores at 6 months are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.039, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 4: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean PCS scores at 1 year are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.278, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 5: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean PCS scores at 2 years are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.804, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test

16. Secondary Outcome: SF-36 Mental Component Summary
Description: The Medical Outcome Study SF-36 Mental Component Summary (MCS) is a subscale of the SF-36 intended to measure mental well-being. It is scored on a scale of 0-100, with higher scores indicating higher levels of well-being.
Time Frame: Baseline, 2 months, 6 months, 1 year, and 2 years post-randomization
Population: Outcomes are analyzed in participants that were alive and completed assessments.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
score on a scale
  Baseline: number analyzed (Participants) | 53 | 59
  Baseline | 47 (1.3) | 48 (1.4)
  2 Months: number analyzed (Participants) | 47 | 51
  2 Months | 49 (1.4) | 50 (1.5)
  6 Months: number analyzed (Participants) | 36 | 46
  6 Months | 50 (1.5) | 48 (1.6)
  1 Year: number analyzed (Participants) | 34 | 39
  1 Year | 50 (1.7) | 46 (2.1)
  2 Years: number analyzed (Participants) | 18 | 30
  2 Years | 52 (1.7) | 50 (1.6)
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean MCS scores at baseline are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.631, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean MCS scores at 2 months are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.759, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 3: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean MCS scores at 6 months are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.391, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 4: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean MCS scores at 1 year are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.222, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 5: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean MCS scores at 2 years are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.527, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test

17. Secondary Outcome: FACT-BMT Score
Description: The Functional Assessment of Cancer Therapy-Bone Marrow Transplant scale (FACT-BMT) is a quality of life instrument that assesses the effects of bone marrow transplantation (BMT) on a patient's physical, social/family, emotional, and functional well-being while taking into consideration BMT-specific concerns. The assessment has 37 questions, each scored on a Likert scale from 0-4. The overall score is computed by adding scores of the questions and falls in the range 0-148, with higher scores indicating higher levels of overall well-being.
Time Frame: Baseline, 2 months, 6 months, 1 year, and 2 years post-randomization
Population: Outcomes are analyzed in participants that were alive and completed assessments.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
Number analyzed (Participants) | 66 | 72
score on a scale
  Baseline: number analyzed (Participants) | 53 | 60
  Baseline | 103 (2.6) | 104 (2.5)
  2 Months: number analyzed (Participants) | 47 | 52
  2 Months | 105 (2.8) | 110 (2.4)
  6 Months: number analyzed (Participants) | 38 | 49
  6 Months | 109 (3.2) | 109 (3.4)
  1 Year: number analyzed (Participants) | 33 | 43
  1 Year | 114 (2.6) | 110 (3.6)
  2 Years: number analyzed (Participants) | 19 | 31
  2 Years | 119 (3.8) | 113 (3.7)
Statistical Analysis 1: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean FACT-BMT scores at baseline are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.763, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 2: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean FACT-BMT scores at 2 months are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.133, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 3: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean FACT-BMT scores at 6 months are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.953, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 4: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean FACT-BMT scores at 1 year are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.398, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test
Statistical Analysis 5: Comparison: Sirolimus, Calcineurin Inhibitor, and Prednisone vs Sirolimus and Prednisone; The null hypothesis is that the mean FACT-BMT scores at 2 years are equal for those receiving either Sirolimus, Calcineurin Inhibitor, and Prednisone or Sirolimus and Prednisone for treatment of chronic GVHD; Test type: Superiority; p = 0.309, t-test, 2 sided — Two-sided testing was performed using a significance level of 0.05; Independent samples t-test

ADVERSE EVENTS:
Time Frame: Three years post-randomization
Arm/Group | Sirolimus, Calcineurin Inhibitor, and Prednisone | Sirolimus and Prednisone
All-Cause Mortality (participants affected / at risk) | 16/66 | 13/72
Serious Adverse Events (participants affected / at risk) | 13/66 | 12/72
Other Adverse Events (participants affected / at risk) | 0/66 | 0/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus, Calcineurin Inhibitor, and Prednisone (N=66) | Sirolimus and Prednisone (N=72)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Splenectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-07-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT01106833/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT01106833/SAP_001.pdf